CLINICAL TRIAL: NCT07321236
Title: Effect of Hands and Feet Exercises on Severity of Taxane-Based Chemotherapy-Induced Peripheral Neuropathy in Patients With Solid Tumors: A Randomized Controlled Trial
Brief Title: Effect of Hands and Feet Exercises on Taxane Based Chemotherapy Induced Peripheral Neuropathy in Patients With Solid Tumors
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Health Sciences Lahore (Other)
Responsible Party: Principal Investigator, Nusrat Hussain, Principal Investigator (MSN student), University of Health Sciences Lahore
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: NHussain
Record Dates: First submitted 2025-12-21; First posted 2026-01-06 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Peripheral Neuropathy
Keywords: Peripheral neuropathy; Taxane; Chemotherapy
MeSH Terms: conditions — Peripheral Nervous System Diseases

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned in a 1:1 ratio to one of two parallel arms and will remain in that assigned arm for the duration of the study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Care (Control) (No Intervention): Standard care
- Hand and Foot Exercise Program + Standard Care (Experimental) (Experimental): Structured Hand and Foot Exercises and standard care
  Interventions: Other: Structured Hand and Foot Exercises

INTERVENTIONS:
Other: Structured Hand and Foot Exercises — The intervention consists of a structured hand and foot exercise program specifically designed for patients experiencing chemotherapy-induced peripheral neuropathy during Taxane-based treatment. It is distinct from general physiotherapy or mobility exercises because it targets peripheral nerve function, joint mobility, and circulation in the hands and feet, aiming to reduce the severity of neuropathic symptoms.
  Arms: Hand and Foot Exercise Program + Standard Care (Experimental)

SUMMARY:
The goal of this clinical trial is to determine whether hand and foot exercises can reduce the severity of Taxane-based chemotherapy-induced peripheral neuropathy (CIPN) in adult cancer patients aged 20-60 years who have Grade 1I neuropathy as defined by the NCI-CTCAE criteria.

The main questions it aims to answer are:

* Do hand and foot exercises reduce the severity of sensory and motor neuropathic symptoms in patients receiving Taxane based chemotherapy?
* Is the severity of peripheral neuropathy lower in the exercise group compared to patients receiving standard care alone? Researchers will compare patients receiving standard care (control group) with those receiving standard care plus a structured hand and foot exercise program (experimental group) to see if the exercises lead to greater improvement in neuropathy severity scores.

Participants will:

* Receive baseline assessment using the EORTC QLQ-CIPN20 questionnaire.
* In the experimental group, learn and perform a 15-minute hand and foot exercise routine on chemotherapy day and continue it at home using a provided brochure.
* Participate in telephonic follow-ups to support compliance and monitor symptoms.
* Undergo a follow-up assessment at alternate week to measure changes in neuropathy severity.

DETAILED DESCRIPTION:
The study focuses on adults between 20 and 60 years old who are receiving Taxane chemotherapy and have early-stage (Grade II) neuropathy. At this stage, patients usually notice changes in sensation, but these changes are still manageable. By starting exercises early, the study aims to see whether regular movement of the hands and feet can help reduce the intensity of these symptoms over time.

Participants will be randomly assigned to one of two groups. One group will continue with their routine medical care for neuropathy, which may include medication and guidance from their healthcare team. The other group will receive the same standard care but will also be taught a short set of hand and foot exercises. These exercises take around 15 minutes to complete and are performed once a day. Patients in the exercise group will first learn the routine on the day of their chemotherapy session and will receive a brochure so they can continue the exercises at home. Telephone check-ins will be used to support patients, answer questions, and encourage regular practice.

To understand how symptoms change, all participants will complete a questionnaire called the EORTC QLQ-CIPN20 at the beginning of the study and again after several weeks. This tool helps measure nerve-related symptoms and how much they affect daily life. The results will allow the research team to compare how symptoms change in both groups over the course of the study.

By examining whether a simple, low-cost exercise routine can make a meaningful difference, this study hopes to offer cancer patients a practical way to manage neuropathy alongside their chemotherapy. If effective, these exercises could become a helpful addition to supportive care in oncology settings, improving comfort and quality of life during treatment.

ELIGIBILITY:
Inclusion Criteria:

* Cancer patients receiving taxane-based chemotherapy on alternate week.
* Age 20-60 years, both male and female.
* Patients having Grade I neuropathy by NCI-CTCEA criteria.

Exclusion criteria:

* Patients with peripheral neuropathy not caused by chemotherapy.

  * Patient with type-1 and type- 2 diabetes.
* Patients with neuropsychiatric disorders.
* Patients having any skin ulcer.
* Individuals having hand foot fracture and varicose veins.
* Individuals with paraplegia.
* Patients receiving radiotherapy.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 58 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2026-08-02 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Severity of peripheral neuropathy | 6 Months
  The primary outcome of this study is the severity of chemotherapy-induced peripheral neuropathy in cancer patients receiving Taxane-based chemotherapy. Severity will be measured using the EORTC QLQ-CIPN20 questionnaire, which assesses sensory symptoms (tingling, numbness, burning), motor symptoms (difficulty gripping or walking), and autonomic symptoms (such as dizziness). Each item is scored from 1 (not at all) to 4 (very much), with higher scores indicating more severe neuropathy. Assessments will be conducted at baseline (week 1) and week 8 to determine whether the hand and foot exercise program reduces symptom severity compared to standard care alone.

CONTACTS AND LOCATIONS:
Overall Officials: Kausar Bano, MBBS, FCPS, Study Chair — Jinnah Hospital,Lahore.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yeo F, Ng CC, Loh KWJ, Molassiotis A, Cheng HL, Au JSK, Leung KT, Li YC, Wong KH, Suen L, Chan CW, Yorke J, Farrell C, Bandla A, Ang E, Lopez V, Sundar R, Chan A. Minimal clinically important difference of the EORTC QLQ-CIPN20 for worsening peripheral neuropathy in patients receiving neurotoxic chemotherapy. Support Care Cancer. 2019 Dec;27(12):4753-4762. doi: 10.1007/s00520-019-04771-8. Epub 2019 Apr 10. PMID 30972646
- See also: Article: "The effect of hand and foot exercises on peripheral neuropathy and quality of life in women with breast cancer: a randomized controlled trial" (2025). — https://link.springer.com/article/10.1007/s00520-025-09145-x
- See also: Article:A Case Study on the Integrated Rehabilitation of Chemotherapy-Induced Peripheral Neuropathy in a Patient with Stage IV Breast Cancer — https://jhrlmc.com/index.php/home/article/view/850
- See also: Article: Striding beyond numbness: a non-randomized controlled study of an exercise program for breast cancer patients with chemotherapy-induced peripheral neuropathy — https://link.springer.com/article/10.1007/s00520-024-09003-2
- Available data/document: Study Protocol — https://jhrlmc.com/index.php/home/article/view/850